CLINICAL TRIAL: NCT02111824
Title: A Multimodality Image-guided System for Peripheral Lung Cancer Diagnosis and Therapy
Acronym: MIMIG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Stephen T. Wong, PhD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00009873; NCT01433822 (obsolete NCT alias)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Lung Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases
Keywords: Lung Cancer; Peripheral lung lesions; Lung biopsy; Minimally invasive; multimodality image-guided intervention system; MIMIG; Indocyanine green; ICG
MeSH Terms: conditions — Lung Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Group 2 (Experimental): During standard of care lung biopsy, the doctor will use the MIMIG system to help guide the needle for the the lung biopsy.
  Interventions: Device: MIMIG System
- Group 3 (Experimental): During standard of care lung biopsy, the doctor will use the MIMIG system to help guide the needle for the lung biopsy. An intravenous (IV) needle placed in the vein to give indocyanine green (IC-Green). Fiber Optic camera will be used to view tissue before biopsy via insertion catheter.
  Interventions: Device: MIMIG System; Drug: Indocyanine Green (ICG)
- Group 1 (No Intervention): Control Group consists of twelve patients who have undergone biopsy of a peripheral lung lesion by using repetitive CT-guidance. Review of medical records only, no further intervention.

INTERVENTIONS:
Device: MIMIG System — Minimally Invasive MultiModality Imaging Guidance System (MIMIG)
  Other Names: Dell Workstation T5500; HP Monitor- LP3065; Aurora Field Generator- A4-00207; Aurora System Control Unit- F4-00275; Aurora Sensor Interface Unit- S4-00556; Introducer Needle- TRAXTAL; Reference- TRAXTAL; Surface Fiducials - Traxtal; Foot Switch- Herge Electric Ltd- 6221-0019
  Arms: Group 2; Group 3
Drug: Indocyanine Green (ICG) — Use of ICG as staining for fiberoptic visualization of lung tissue via introducer needle prior to obtaining tissue samples.
  Other Names: indocyanine green (IC-Green).; 3 mg/kg by vein before lung biopsy.; Indocyanine green; IC-Green; ICG
  Arms: Group 3

SUMMARY:
The goal of this clinical research study is to test the use of a minimally invasive multimodality image-guided (MIMIG) intervention system used for performing a lung biopsy. The safety of the MIMIG intervention system will also be studied.

DETAILED DESCRIPTION:
Group 2:

If the patient agrees to take part in this study, the following information about their routine standard of care lung biopsy will be collected:

The accuracy of the procedure How long it takes to complete the procedure How long the needle is inserted to collect the biopsy sample The number of CT scans used during the procedure The radiation dose level used Any complications and/or side effects the patient may experience The results of the diagnosis from the biopsy sample Researchers will take appropriate steps to keep the patient's information private. However, there is no guarantee of absolute privacy. The patient's information will be kept in a password-protected computer at MD Anderson for up to 7 years and will only be permitted to be viewed by the study doctor and members of the research staff.

During the patient's routine lung biopsy, the doctor will use the MIMIG intervention system to help guide the needle for the biopsy the lung biopsy.

Length of Study:

The patient's active participation on this study will be over after the lung biopsy procedure is over.

Description of Procedure:

The first CT scan will be used as a map to guide a needle into the tumor with the MIMIG intervention system. After that, a second CT scan will be done to confirm that the needle tip has been properly inserted inside the lung tumor. Based on the results from these images, the tumor will then be biopsied the same way it would be as part of normal routine care.

This is an investigational study. The use of the MIMIG intervention system to help guide the needle for the lung biopsy is not FDA approved or commercially available. The use of the MIMIG intervention system is investigational.

Up to 24 patients will take part in this study. All will be enrolled at MD Anderson.

Group 3:

If the patient agrees to take part in this study, the following information about the patient's routine standard of care lung biopsy will be collected:

The accuracy of the procedure How long it takes to complete the procedure How long the needle is inserted to collect the biopsy sample The number of CT scans used during the procedure The radiation dose level used Any complications and/or side effects the patient may experience The results of the diagnosis from the biopsy sample Researchers will take appropriate steps to keep the patient's information private. However, there is no guarantee of absolute privacy. The patient's information will be kept in a password-protected computer at MD Anderson and will only be permitted to be viewed by the study doctor and members of the research staff.

During the patient's routine lung biopsy, the doctor will use the MIMIG intervention system to help guide the needle for the biopsy the lung biopsy. The patient will also have an intravenous (IV) needle placed in the patient's vein to give the patient indocyanine green (IC-Green). IC-Green is a dye that allows researchers to see the patient's veins and other organs during the biopsy.

Length of Study:

After the lung biopsy is complete, the patient's active participation on this study will be over.

Description of Procedure:

The first CT scan will be used as a map to guide a needle into the tumor with the MIMIG intervention system. After that, a second CT scan will be done to confirm that the needle tip has been properly inserted inside the lung tumor. A fiberoptic endoscope (a small camera with a light) will be inserted through the CT guided needle to the tumor to help doctors see the tumor blood vessels. IC-Green will also be given by IV to allow doctors to see the blood vessels of the tumor. Based on the results from these images, the tumor will then be biopsied the same way it would be as part of normal routine care.

This is an investigational study. The use of the MIMIG intervention system to help guide the needle for the lung biopsy is not FDA approved or commercially available. The use of the MIMIG intervention system is investigational. The use of fiberoptic endoscope for lung tumor vessels imaging is not FDA approved or commercially available. The use of fiberoptic endoscope is investigational. The use of IC-Green in combination with fiberoptic endoscope for lung tumor vessels imaging is not FDA approved or commercially available. The use of IC-Green in combination with fiberoptic endoscope is investigational.

Up to 24 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years) subjects with peripheral lung lesions that are <1.5 cm in size who are planning to undergo percutaneous image guided lung biopsy as part of their routine medical care.
* 2. Ability to understand and willingness to sign Informed Consent Document (ICD)

Exclusion Criteria:

* Age less than 18 years.
* Pregnant or nursing females.
* Known allergy to iodine or intravenous contrast agent.
* Known allergy or anaphylactic reaction to indocyanine green (ICG).
* Patients with renal dysfunction (GFR <60) or patients on dialysis
* Patients with liver dysfunction: total bilirubin > 2.5 mg/dl; albumin < 2.5 mg/dl; alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 5 times upper limits of normal
* Uncorrectable coagulopathy prohibiting biopsy. (INR > 1.5 and/ or platelets < 50,000)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Technical Success Rate of Biopsy Using the MIMIG system With + Without Fiber-Optical Imaging | 3 Mos
  Technical success rate of completing the biopsy procedure using the MIMIG system with and without fiber-optical imaging measured where technical success is defined as the ability to use the navigational components of the MIMIG system to obtain a tissue specimen from a lung nodule; ability to use the navigational components of the system during the biopsy procedure, the ability to successfully perform optical imaging of the lung nodule and the ability to obtain a tissue specimen from the lung nodule.

CONTACTS AND LOCATIONS:
Overall Officials: Alda Tam, MD, Principal Investigator — MD Anderson Cancer Center Interventional Radiology
Locations (1):
- MD Anderson Cancer Center Interventional Radiology Dept., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No